CLINICAL TRIAL: NCT04435886
Title: A 12-weeks Prospective, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of a Probiotic in the Treatment of Fibromyalgia
Brief Title: Use of a Probiotic in the Treatment of Fibromyalgia (FIBROPROB)
Acronym: FIBROPROB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biopolis S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIBRO.PROB
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-06

CONDITIONS: Fibromyalgia
Keywords: Probiotic; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: 12-week randomized, double-blind, parallel-group, placebo-controlled study
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): A multi-strain probiotic
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Identical placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Probiotic mixture with maltodextrin as a carrier.
  Arms: Probiotic group
Dietary Supplement: Placebo — Placebo comparator with maltodextrin as a carrier.
  Arms: Placebo group

SUMMARY:
This study aims to understand the efficacy of two probiotic interventions as prophylaxes of fibromyalgia symptoms in individuals diagnosed.

The primary outcome measure will be the progression and treatment of fibromyalgia, defined as a decrease in the Fibromyalgia Impact Questionnaire (FIQ) score, other otucomes will be the effect on the symptoms of anxiety and depression associated with fibromyalgia, defined as a decrease in the Hospital Anxiety and Depression Scale (HAD) score; perception of pain by scoring on a Visual Analogical Pain Scale (VAS), and differences in the patient's usual medical treatment. Finally adverse effects will be evaluated.

The study will have two arms: one arm including a probiotic preparation and a placebo arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 - 65 years.
2. Signature of informed consent by the patient.
3. Patients diagnosed according to the 2010 American College of Rheumatology (ACR) diagnostic criteria for fibromyalgia

Exclusion Criteria:

11. Women who are pregnant, breastfeeding or who do not commit to using an effective method of contraception during the course of the study.

2. Known allergy to any of the components of the study product or the placebo. 3. Consumption of antibiotics in the 2 weeks prior to the start of the study. 4. Consumption of probiotics in the 2 months prior to the start of the study. 5. Evidence of neuropsychiatric disorders including: Parkinson's disease, psychotic disorder, bipolar depression 6. Regular consumption of alcohol in excess of 45 g ethanol/day in the year prior to study inclusion.

7. Any concurrent malignant pathology known at the time of inclusion in the study or serious metabolic, cardiovascular, renal, hepatic or gastrointestinal diseases which may lead to non-completion of the study according to the investigator's criteria.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-02-02 (Estimated); Study Completion 2021-05-02 (Estimated)

PRIMARY OUTCOMES:
Score on the Fibromyalgia Impact Questionnaire (FIQ) | 4-week
  Score on the Fibromyalgia Impact Questionnaire (FIQ) in weeks 4
Score on the Fibromyalgia Impact Questionnaire (FIQ) | 8-week
  Score on the Fibromyalgia Impact Questionnaire (FIQ), The score range is form 0 to 100, where each question has an score from 0 to 10. Higher scores refers a higher impact of fybromialgia in lifestile where 0 is the best functional capacity and higher quality of life and 100 the worst stat, in weeks 8
Score on the Fibromyalgia Impact Questionnaire (FIQ) | 12-week
  Score on the Fibromyalgia Impact Questionnaire (FIQ), The score range is form 0 to 100, where each question has an score from 0 to 10. Higher scores refers a higher impact of fybromialgia in lifestile where 0 is the best functional capacity and higher quality of life and 100 the worst stat, in weeks 12.

SECONDARY OUTCOMES:
Score on the Hospital Anxiety and Depression Scale (HAD) | 4 weeks
  Score on the Hospital Anxiety and Depression Scale (HAD), To determine the levels of anxiety and depression that a person is experiencing. It is a fourteen item scale; seven items are related to anxiety and seven to depression. Each item is scored from 0-3, being the total score from 0 to 21 for either anxiety or depression. The higher score the worse state. in weeks 4
Score on the Hospital Anxiety and Depression Scale (HAD) | 8 weeks
  Score on the Hospital Anxiety and Depression Scale (HAD), To determine the levels of anxiety and depression that a person is experiencing. It is a fourteen item scale; seven items are related to anxiety and seven to depression. Each item is scored from 0-3, being the total score from 0 to 21 for either anxiety or depression. The higher score the worse state. In weeks 8
Score on the Hospital Anxiety and Depression Scale (HAD) | 12 weeks
  Score on the Hospital Anxiety and Depression Scale (HAD), To determine the levels of anxiety and depression that a person is experiencing. It is a fourteen item scale; seven items are related to anxiety and seven to depression. Each item is scored from 0-3, being the total score from 0 to 21 for either anxiety or depression. The higher score the worse state. In weeks 12.
Visual Analogical Pain Scale (VAS) Score | 12 weeks
  Visual Analogical Pain Scale (VAS) Score. It is a unidimensional continuous measure of pain intensity. It comprises a horizontal (HVAS) or vertical (VVAS) line, 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme. For pain intensity, the scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]). in weeks 12
Changes to a patient's usual medical treatment for fibromyalgia | 4 weeks
  Changes to a patient's usual medical treatment for fibromyalgia, in weeks 4 Little or no impact (46 or less) Some impact (50 -55) Substantial impact (56-59) Severe impact (60-78)
Changes to a patient's usual medical treatment for fibromyalgia | 8 weeks
  Changes to a patient's usual medical treatment for fibromyalgia, in weeks 8 Little or no impact (46 or less) Some impact (50 -55) Substantial impact (56-59) Severe impact (60-78)
Changes to a patient's usual medical treatment for fibromyalgia | 12 weeks
  Changes to a patient's usual medical treatment for fibromyalgia, in weeks 12 Little or no impact (46 or less) Some impact (50 -55) Substantial impact (56-59) Severe impact (60-78)
Treatment adherence rate | 4 weeks
  Treatment adherence rate using the returned capsules, in weeks 4
Treatment adherence rate | 8 weeks
  Treatment adherence rate using the returned capsules, in weeks 8
Treatment adherence rate | 12 weeks
  Treatment adherence rate using the returned capsules, in weeks 12
Number of adverse events | 4 weeks
  Numbre od adverse effects reported, 4 weeks
Number of adverse events | 8 weeks
  Numbre od adverse effects reported, 8 weeks
Number of adverse events | 12 weeks
  Numbre od adverse effects reported, 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Vinalopó, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No